CLINICAL TRIAL: NCT01187420
Title: Real Time Monitoring for Cerebral Vasospasm Using Bilateral Processed Electroencephalogram (EEG)
Brief Title: Bilateral Bispectral Index (BIS) Study
Acronym: BIS
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0470
Record Dates: First submitted 2010-03-31; First posted 2010-08-24 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Cerebral Vasospasm; Delayed Cerebral Ischemia; Subarachnoid Hemorrhage
Keywords: Cerebral vasospasm; delayed cerebral ischemia (DCI); subarachnoid hemorrhage (SAH) patients
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EEG and Cerebral Vasospasm: Cerebral Vasospasm and role of BIS vista monitor in Subarachnoid Hemorrhage (SAH) patients

SUMMARY:
The purpose of this study is to assess real time changes in raw and processed EEG in relation to the clinical and radiological evidence of cerebral vasospasm.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) is a prevalent and morbid condition (45%-30 day mortality). One of the major causes of reduced cerebral blood flow (CBF) after initial SAH is cerebral vasospasm. Early treatment of cerebral vasospasm (< 2 hr) is necessary for improved neurologic outcome. Hence, there is significant interest in development of a monitor. The most common bedside diagnostic tool is Transcranial Doppler (TCD) which is controversial given its low sensitivity and specificity. TCD is not a continuous monitor and is user dependent. Many centers rely on Cerebral Angiography for diagnosis of vasospasm; however angiographic spasm does not correlate with outcome. EEG can detect changes in cerebral blood flow which precede clinical decline but is technically difficult to perform and not practical for continuous monitoring.

Processed EEG monitors have become somewhat popular in the operating setting for assessment of depth of anesthesia. The recent introduction of bilateral 4 channel disposable probes presents to opportunity to use EEG as a non-invasive continuous monitor for vasospasm. We propose a prospective observational study to assess real time changes in raw and processed EEG which we will correlate with clinical and radiologic evidence of vasospasm. Our primary clinical endpoint will be the determination of delayed cerebral ischemia. This modality could prove to be a significant clinical advantage for patients suffering from SAH.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women of any age and ethnicity within 48 hours of subarachnoid hemorrhage (SAH)

Exclusion Criteria:

* Age < 18 years
* Greater than 48 hours past the initial hemorrhage
* Previous history of stroke of any etiology
* Inability to consent for themselves or have a proxy to consent for them (implied consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurosurgical ICU patients with Subarachnoid Hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Detection of delayed cerebral ischemia (DCI) utilizing Bispectral Index (BIS) | 10 days stay at the NSICU

SECONDARY OUTCOMES:
BIS correlation with angiography and transcranial doppler flow for detection of cerebral vasospasm | 10 days stay at the NSICU

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Deiner, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Cross DT 3rd, Tirschwell DL, Clark MA, Tuden D, Derdeyn CP, Moran CJ, Dacey RG Jr. Mortality rates after subarachnoid hemorrhage: variations according to hospital case volume in 18 states. J Neurosurg. 2003 Nov;99(5):810-7. doi: 10.3171/jns.2003.99.5.0810. PMID 14609158
- [Background] Broderick JP, Brott TG, Duldner JE, Tomsick T, Leach A. Initial and recurrent bleeding are the major causes of death following subarachnoid hemorrhage. Stroke. 1994 Jul;25(7):1342-7. doi: 10.1161/01.str.25.7.1342. PMID 8023347
- [Background] Sehba FA, Bederson JB. Mechanisms of acute brain injury after subarachnoid hemorrhage. Neurol Res. 2006 Jun;28(4):381-98. doi: 10.1179/016164106X114991. PMID 16759442
- [Background] Heros RC, Zervas NT, Varsos V. Cerebral vasospasm after subarachnoid hemorrhage: an update. Ann Neurol. 1983 Dec;14(6):599-608. doi: 10.1002/ana.410140602. PMID 6651248
- [Background] Claassen J, Hirsch LJ, Kreiter KT, Du EY, Connolly ES, Emerson RG, Mayer SA. Quantitative continuous EEG for detecting delayed cerebral ischemia in patients with poor-grade subarachnoid hemorrhage. Clin Neurophysiol. 2004 Dec;115(12):2699-710. doi: 10.1016/j.clinph.2004.06.017. PMID 15546778
- [Background] Aaslid R, Huber P, Nornes H. Evaluation of cerebrovascular spasm with transcranial Doppler ultrasound. J Neurosurg. 1984 Jan;60(1):37-41. doi: 10.3171/jns.1984.60.1.0037. PMID 6689726
- [Background] Lysakowski C, Walder B, Costanza MC, Tramer MR. Transcranial Doppler versus angiography in patients with vasospasm due to a ruptured cerebral aneurysm: A systematic review. Stroke. 2001 Oct;32(10):2292-8. doi: 10.1161/hs1001.097108. PMID 11588316
- [Background] Claassen J, Bernardini GL, Kreiter K, Bates J, Du YE, Copeland D, Connolly ES, Mayer SA. Effect of cisternal and ventricular blood on risk of delayed cerebral ischemia after subarachnoid hemorrhage: the Fisher scale revisited. Stroke. 2001 Sep;32(9):2012-20. doi: 10.1161/hs0901.095677. PMID 11546890
- [Background] Frontera JA, Fernandez A, Schmidt JM, Claassen J, Wartenberg KE, Badjatia N, Connolly ES, Mayer SA. Defining vasospasm after subarachnoid hemorrhage: what is the most clinically relevant definition? Stroke. 2009 Jun;40(6):1963-8. doi: 10.1161/STROKEAHA.108.544700. Epub 2009 Apr 9. PMID 19359629
- [Background] Rosenwasser RH, Armonda RA, Thomas JE, Benitez RP, Gannon PM, Harrop J. Therapeutic modalities for the management of cerebral vasospasm: timing of endovascular options. Neurosurgery. 1999 May;44(5):975-9; discussion 979-80. doi: 10.1097/00006123-199905000-00022. PMID 10232530
- [Background] Sen I, Puri GD, Bapuraj JR. Early detection of cerebral vasospasm during a neurointerventional procedure using the BIS. Anaesth Intensive Care. 2005 Oct;33(5):691-2. No abstract available. PMID 16235500
- [Background] Claassen J, Mayer SA, Hirsch LJ. Continuous EEG monitoring in patients with subarachnoid hemorrhage. J Clin Neurophysiol. 2005 Apr;22(2):92-8. doi: 10.1097/01.wnp.0000145006.02048.3a. PMID 15805808
- [Background] Towle VL, Bolanos J, Suarez D, Tan K, Grzeszczuk R, Levin DN, Cakmur R, Frank SA, Spire JP. The spatial location of EEG electrodes: locating the best-fitting sphere relative to cortical anatomy. Electroencephalogr Clin Neurophysiol. 1993 Jan;86(1):1-6. doi: 10.1016/0013-4694(93)90061-y. PMID 7678386
- [Background] Vespa PM, Nuwer MR, Juhasz C, Alexander M, Nenov V, Martin N, Becker DP. Early detection of vasospasm after acute subarachnoid hemorrhage using continuous EEG ICU monitoring. Electroencephalogr Clin Neurophysiol. 1997 Dec;103(6):607-15. doi: 10.1016/s0013-4694(97)00071-0. PMID 9546487
- [Background] Labar DR, Fisch BJ, Pedley TA, Fink ME, Solomon RA. Quantitative EEG monitoring for patients with subarachnoid hemorrhage. Electroencephalogr Clin Neurophysiol. 1991 May;78(5):325-32. doi: 10.1016/0013-4694(91)90094-k. PMID 1711451
- [Background] Schultz A, Siedenberg M, Grouven U, Kneif T, Schultz B. Comparison of Narcotrend Index, Bispectral Index, spectral and entropy parameters during induction of propofol-remifentanil anaesthesia. J Clin Monit Comput. 2008 Apr;22(2):103-11. doi: 10.1007/s10877-008-9111-6. Epub 2008 Feb 21. PMID 18288579